CLINICAL TRIAL: NCT01703442
Title: Perioperative Relevance of Intraoperative Anuric Episodes Within a Goal-directed Haemodynamic Algorithm in Patients Undergoing Laparotomy Due to Epithelial Ovarian Cancer
Brief Title: Intraoperative Anuric Episodes in Patients Undergoing Laparotomy
Status: Withdrawn | Type: Observational
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: EPERIA
Record Dates: First submitted 2012-09-24; First posted 2012-10-10 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Intraoperative Anuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ovarian cancer patients: Perioperative primary epithelial ovarian cancer patients

SUMMARY:
A single-center prospective observational study. This study examines urine flow and haemodynamic parameters during abdominal surgery and analyses the association to postoperative renal function and markers and to postoperative clinical outcome.

Primary hypothesis:

• Within a goal-directed haemodynamic protocol during gynecologic cancer surgery there are phases of temporary anuria.

Secondary hypothesis:

* Perioperative anuric phases are directly associated to the postoperative increase of NGAL (neutrophil gelatinase-associated lipocalin) and creatinine
* Perioperative renal dysfunction is directly associated to postoperative complications and functional recovery of patients
* A response of urine flow to a standardized postoperative diuretic bolus can identify patients who benefit from a pharmaceutical fluid mobilization
* Within a goal-directed haemodynamic protocol during gynaecologic cancer surgery, the methods for the measurement of stroke volume of the heart differ

ELIGIBILITY:
Inclusion Criteria:

* Offered patient information and written informed consent
* Female patients aged greater than or equal to 18 years for cytoreductive surgery of a primary epithelial ovarian tumour

Exclusion Criteria:

* Patients with relapse Ovarian Cancer
* Patients aged less than 18 years
* Persons without the capacity to consent
* Unability of German language use
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* (Unclear) history of alcohol or substances disabuse
* Coworker of the Charité
* Advanced disease of the oesophagus or upper respiratory tract at the beginning of hospitalisation
* Operation in the area of the oesophagus or nasopharynx within the last two months before participation in the study
* Neurological or psychiatric disease at the beginning of hospitalisation
* CHF (congestive heart failure) according to (New York Heart Association) classification - NYHA class IV at the beginning of hospitalisation
* American Society of Anaesthesiologists (ASA) classification greater than IV
* Renal insufficiency (dependency of haemodialysis) at the beginning of hospitalisation
* Pulmonal oedema in thorax x-ray at the beginning of hospitalisation
* History of intracranial hemorrhage within one year before participation in the study
* Conditions following venous thrombosis within the last three years before study inclusion
* Known allergies or hypersensitivity on colloidal, starch or gelatine infusion solutions
* Diabetes mellitus with signs of severe neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients being treated in the Department of Gynecology and Obstetrics, Campus Virchow Klinikum, Charité - Universitaetsmedizin Berlin.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Exact measurement of urine production | During the operation and in the 72-hour postoperative sample period
  Exact measurement of urine production (number of anuric episodes anf duration of anuric episodes in minutes)

SECONDARY OUTCOMES:
Exact measurement of urine production | During the operation and in the 72-hour postoperative sample period
  Exact measurement of urine production (amount in milliliter)
Biomarker for renal injury, Neutrophil gelatinase-associated lipocalin (NGAL) and creatinine | During the operation and in the 72-hour postoperative sample period
  Parameters from blood sample
Hemodynamic parameters | During the operation
Blood loss | During the operation
Depth of Anesthesia | During the operation
  Measuring depth of Anesthesia by Bispectral Index Monitoring
Organ dysfunctions | During the operation and in the 72-hour postoperative sample period
Postoperative pain | In the 72-hour postoperative sample period
Body weight development | In the 72-hour postoperative sample period
Duration until fulfilment of hospital discharge criteria | Participants will be followed for the duration of an expected average of 4 weeks
ICU and hospital length of stay | Participants will be followed for the duration of intensive care unit stay and hospital stay, an expected average of 4 weeks
Quality of life and functional status | Participants will be followed for the duration of hospital stay, an exspected average of 4 weeks
Inflammatory parameters | In the 72-hour postoperative sample period
Amount of vasopressors | During the operation and in the 72-hour postoperative sample period

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum, Charité - Universitaetsmedizin, Berlin, State of Berlin, Germany